CLINICAL TRIAL: NCT00102895
Title: An Open-Label, Multi-Center, Phase 2 Study Of Cp 724,714 In Patients With Her2 Overexpressing Metastatic Breast Cancer That Has Progressed After Chemotherapy For Metastatic Disease And Is Previously Untreated With A Her2 Inhibitor
Brief Title: A Research Study of CP-724,714 in Patients With HER2 Overexpressing Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See Detailed Description
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4031003
Record Dates: First submitted 2005-02-03; First posted 2005-02-04 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-08

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — 2-methoxy-N-(3-(4-((3-methyl-4-((6-methyl-3-pyridinyl)oxy)phenyl)amino)-6-quinazolinyl)-2-propenyl)acetamide

INTERVENTIONS:
Drug: CP-724,714

SUMMARY:
The main purpose of this research study is to see if the study drug, named CP-724,714, can help in the treatment of certain breast cancers that have spread to other locations in the body. Other goals of this study are to measure how long it may take for the cancer to get worse (progress), to see if there are any side effects from the study drug, to check the amount of study drug in the blood at different times, and to check to see if there is any relationship between certain blood tests and how patients may respond to the study drug.

About 25 subjects at 4 sites (hospitals and clinics) in Bulgaria and Russia will be involved in the trial. Participation in this study can last up to 48 weeks, depending on the participant's toleration of the study drug and the response of her tumor(s) to the study drug. All participants will receive CP-724,714, at a daily dose of 250 mg (4 pills) every 12 hours.

DETAILED DESCRIPTION:
Pfizer decided to terminate clinical protocol A4031003 on October 7, 2005 due to the excessive number of patients with grade 3 liver function test elevations and lack of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Signed written and voluntary informed consent
* Histologically or cytologically confirmed breast cancer
* Stage IV (metastatic) breast cancer
* Biopsy (fresh or archival) of primary breast cancer or metastatic site demonstrating HER2 gene amplification as determined in study-specified central laboratory by fluorescence in situ hybridization (FISH)
* Prior treatment and progressive disease with at least 1 but not more than 2 cytotoxic chemotherapy regimen(s) for metastatic disease
* Those for whom the use of an investigational HER2 inhibitor is appropriate because they do not have access to approved HER2 inhibitors (e.g., Herceptin®) or for whom treatment with currently available HER2 inhibitors is inappropriate
* Limited visceral disease burden (i.e., <30% involvement of any organ) and limited disease-related symptoms (i.e., well controlled with supportive care measures)
* Presence of at least one measurable target lesion [i.e., malignant tumor mass that can be accurately measured in at least 1 dimension of >=2 cm with conventional radiographic techniques or magnetic resonance imaging, or >=1 cm with spiral CT scan as per RECIST], excluding previously irradiated lesions, bone metastasis or pleural effusion as sole manifestations of disease. If the measurable disease is restricted to a solitary lesion, its neoplastic nature must be confirmed by cytology/histology
* Eastern Cooperative Oncology Group (ECOG) performance status 0 1
* Patient available for treatment, monitoring, and follow-up. Willing and able to comply with scheduled visits, therapy plan, laboratory tests and blood sampling for pharmacokinetic (PK) analyses
* Recovery to baseline or NCI CTCAE Version 3.0 Grade 1 toxicity from all acute effects related to prior treatment, except alopecia
* Adequate Bone Marrow Function, including: a. Absolute neutrophil count (ANC) >=1500 cells/mm3; b. Platelets >=100,000 cells/mm3
* Adequate Renal Function, including: a. Estimated creatinine clearance >=60 mL/min; b. SrCr <1.5 x ULN
* Adequate Liver Function, including: a. Bilirubin <=ULN (upper limit of normal); b. AST (SGOT) <=2.5 x ULN; c. ALT (SGPT) <=2.5 x ULN
* Adequate Cardiac Function, including: a. 12-Lead electrocardiogram (ECG) with normal tracing or non clinically significant changes that do not require medical intervention; b. QTc interval <=450 msec and without history of Torsades des Pointes or other symptomatic QTc abnormality; c. Left ventricular ejection fraction (LVEF) >= institutional lower limit of normal and 45% as measured by echocardiogram or multi gated radionuclide angiography (MUGA) within 4 weeks prior to start of study treatment
* >= 18 years old
* Female

Exclusion Criteria:

* Women of child-bearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and up to 4 weeks after study
* Women who are pregnant or breastfeeding
* Women with a positive pregnancy test on enrollment or within 72 hours prior to study drug administration
* Prior treatment with trastuzumab (Herceptin®) or other HER2-targeting agents [e.g., lapatinib (GW572016), pertuzumab (Omnitarg™; rhuMab 2C4), CI 1033, EKB 569, CP 724,714]
* Cumulative dose >450 mg/m2 of doxorubicin or doxorubicin equivalents
* Prior high-dose chemotherapy requiring hematopoetic stem cell transplantation within 12 months of study treatment start
* Radiotherapy, investigational chemotherapy, biologic therapy within 4 weeks of study treatment start
* Previous (within the last 5 years) or current malignancies arising from sites other than breast, except for adequately treated basal cell or squamous cell skin cancer or in situ carcinoma of the cervix uteri
* Known or clinically suspected brain metastasis or leptomeningeal disease (no screening CT scan required) requiring therapy. Patients with asymptomatic previously treated CNS metastases that no longer require therapy or corticosteroids/anticonvulsants for at least 4 weeks prior to start of study treatment are eligible
* Any clinically significant gastrointestinal abnormalities, which may impair intake, transit or absorption of the study drug, such as the inability to take oral medication in tablet form, prior complete/partial gastrectomy or intestinal resection, or a requirement for H2 antagonists or proton pump inhibitors
* Any mental disorder that would limit the understanding or rendering of informed consent and/or compromise compliance with the requirements of this protocol
* Uncontrolled or significant cardiovascular disease, including: a. Myocardial infarction within 12 months; b. Uncontrolled angina within 6 months; c. Congestive heart failure within 6 months or left ventricular ejection fraction below local institutional lower limit of normal or below 45%; d. Diagnosed or suspected congenital long QT syndrome; e. Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsade de pointes); f. Prolonged QTc interval on pre-entry electrocardiogram (>450 msec); g. Any history of second or third degree heart block (may be eligible if currently have a pacemaker); h. Heart rate <50/minute on pre-entry electrocardiogram; i. Uncontrolled hypertension
* History of drug-induced hyperbilirubinemia
* Concurrent treatment with approved or investigational chemotherapy, hormonal therapy, immunotherapy, or radiotherapy (hormone replacement therapy is permitted)
* Concurrent treatment with H2 antagonists and/or proton pump inhibitors. However, H2 antagonists can be used for the treatment of an unexpected hypersensitivity reaction during the study period. Antacids are allowed but only up to 2 hours before and 2 hours after study drug administration
* Concurrent treatment or treatment within 4 weeks of first dose with potent and/or irreversible CYP3A4 inhibitors including: ketoconazole, itraconazole, troleandomycin, clarithromycin, erythromycin, ritonavir, indinavir, nelfinavir, saquinavir, nefazodone, mibefradil, amiodarone and grapefruit juice
* Concurrent treatment or treatment within 4 weeks of first dose with potent inducers of CYP3A4 including: rifampin, rifabutin, rifamycins, phenytoin, barbiturates, carbamazepine, glucocorticoids, modafinil, phenobarbital, troglitazone, pioglitazone, efavirenz, nevirapine, dexamethasone, and St. John's wort
* Prisoners or patients who are compulsorily detained or involuntarily incarcerated (e.g., for treatment of infectious disease, psychiatric illness, etc.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2005-04; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Tumor Response

SECONDARY OUTCOMES:
Safety/Tolerability and Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer